CLINICAL TRIAL: NCT03590197
Title: Effect of Melatonin on Seizure Outcome, Neuronal Damage and Quality of Life in Patients With Generalized Epilepsy: A Randomized, add-on Placebo-controlled Clinical Trial
Brief Title: Effect of Melatonin on Seizure Outcome, Neuronal Damage and Quality of Life in Patients With Generalized Epilepsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, RITUPARNA MAITI, Additional professor, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IEC/AIIMSBBSR/PGTh/18-19/02
Record Dates: First submitted 2018-07-06; First posted 2018-07-18 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Generalized Epilepsy
Keywords: Melatonin; Neuron-specific Enolase; Responder rate
MeSH Terms: conditions — Epilepsy, Generalized | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The recruited patients will be randomized by simple randomization into two treatment groups using computer-generated random codes. The random allocation code of the participants will be generated by PI who will not be involved in the patient recruitment. The codes will be assigned to a sequence of numbers and the numbered stickers will be pasted on the similar looking drug containers. The drug containers will be given to another investigator who will be responsible for patient recruitment. This process ensured allocation concealment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Arm (Placebo Comparator): The patients in Control Arm will receive placebo with valproate (20 mg/kg).
  Interventions: Other: Placebo
- Melatonin Arm (Experimental): The Experimental Arm will receive tablet melatonin as an add-on to valproate. Melatonin will be prescribed 3 mg/day to the patients and will be advised to take 30 minutes before bedtime.
  Interventions: Drug: Melatonin 3 mg

INTERVENTIONS:
Drug: Melatonin 3 mg — Melatonin 3 mg/ day with Valproate
  Arms: Melatonin Arm
Other: Placebo — Placebo with Valproate
  Arms: Control Arm

SUMMARY:
Epilepsy is one of the most common and frequently encountered neurological conditions that impose a huge burden on the healthcare systems. Despite the abundance of antiepileptic drugs (AEDs) available, 30% of people continue to have seizures even after long-term therapy of 6-8 years. This group of people requires a more aggressive treatment since monotherapy, the first choice scheme, is not sufficient to control seizure and its complications, multiple drug therapy or polytherapy often results in the culmination of unwanted effects. The need for an add-on AEDs with a good safety profile is of utmost importance.The beneficial effects of melatonin on sleep, its wide safety window, and its ability to cross the blood-brain barrier have the potential to improve the quality of life in seizure patients. Various animal studies have suggested that melatonin receptors are the potential targets for anticonvulsant drug development. In animal studies, melatonin was found to suppress generalized seizure and seizure susceptibility and it also has neuroprotection and synapse modulating properties. Some clinical trials mostly on paediatric population also found that melatonin can improve the clinical outcome in epilepsy. Therefore, we have planned to conduct a randomized, add-on placebo-controlled clinical trial on the effect of melatonin on seizure outcome, neuronal damage and quality of life in adult patients with generalized seizure.

DETAILED DESCRIPTION:
Epilepsy is a chronic disabling neurologic condition which often leads to numerous adverse long-term neurologic complications, such as behavioural and cognitive deficits, increased susceptibility to recurrent seizures, and neuronal injury or death. Cognitive dysfunction, depression, anxiety and sleep disorders are some of the highly prevalent and most debilitating complications of epilepsy. Despite the abundance of antiepileptic drugs (AEDs), even after long-term treatment of 6-8 years, 30% of patients continue having seizures. This group of patients requires a more aggressive treatment, since monotherapy fails to control seizures, considering the fact that the number of seizures is the single most important predictive factor for both early and long-term remission of seizures. Nevertheless, polytherapy often results in a number of adverse effects. The need for better-tolerated add-on therapy is the need of the hour to overcome this therapeutic hurdle.

Melatonin, an endogenous hormone, acting through MT1 and MT2 receptors exert a depressive effect on brain excitability and have been shown to exert an anticonvulsant activity in various animal models. In some clinical trials also it has been found that add-on melatonin therapy improves the clinical outcome. Uberoset al evaluated the sleep-wake pattern, plasma melatonin levels and the urinary excretion of its metabolite among children with severe epileptic disorders, before and after a therapeutic trial with melatonin. They found sleep efficiency was significantly higher and better controls of convulsive episodes were achieved with among patients who received melatonin. Goldberg-Stern et aland Elkhayat et al concluded that melatonin could be effective and safe for decreasing seizure frequency and severity in patients with intractable epilepsy. Gupta et al found that melatonin has the potential to improve quality of life in pediatric epilepsy because of its beneficial effects on sleep, its wide safety window, and its ability to cross the blood-brain barrier. In another study by Jain SV et al melatonin resulted in a statistically significant decrease in sleep onset latency and wakefulness after sleep onset. Guptaet al also concluded that add-on melatonin can be of promise in the pharmacotherapy of pediatric epilepsy and as an adjunct, can be a putative neuroprotector in conditions involving oxidative stress like epilepsies. Dabak et al and Brazil et measured melatonin in febrile seizure and temporal lobe epilepsy and found to be lower in epilepsy in comparison to the controls.

Our literature review reveals that till date most of the clinical studies on the effect of melatonin in epilepsy have been conducted in the pediatric population and there is no clinical trial done on its effect on seizure outcome, neuroprotective effect, sleep and circadian rhythm and quality of life in adult patients with epilepsy. So the present randomized clinical trial has been designed to fill the knowledge gap and evaluate the effect of add-on melatonin on seizure severity, neuronal damage and sleep quality in adult patients suffering from a generalized seizure.

ELIGIBILITY:
Inclusion Criteria:

* All patients with the clinical diagnosis of generalized epilepsy with generalised onset motor seizure (ILAE 2017) with a history of an episode of seizure within 72 hours of presentation.
* Patients aged 18-60 years, of either sex.
* Treatment-naive patients or patients who had not taken any treatment for at least 4 weeks before inclusion.

Exclusion Criteria:

* History of any recent traumatic brain injury, cerebral ischemia/TIA/stroke.
* Patients with neuroendocrinal tumors.
* History of any invasive neurosurgical/non-invasive neuropsychiatric procedure.
* Patients who are already under treatment for the presenting conditions.
* Medication history of psychoactive or central nervous system depressant drugs.
* Pregnant and nursing women.
* Patients with a history of allergy to valproate, melatonin or other melatonin agonists.
* Patients with drug/alcohol abuse.
* Patients with any hepatic dysfunction.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-04-12 (Actual)

PRIMARY OUTCOMES:
Change in Responder Rate from baseline | Baseline, 8 weeks
  Responder rate is defined as percentage of patients having ≥50% reduction in seizure frequency.

SECONDARY OUTCOMES:
Change in seizure severity from baseline | Baseline , 8 weeks
  The change in seizure severity in terms of change in Chalfont-National Hospital seizure severity scale (NHS3)
Change in neuronal damage from baseline | Baseline, 8 weeks
  The change in neuronal damage in terms of change in serum NSE (Neuron-specific Enolase) level
Change in sleep quality from the baseline | Baseline, 8 weeks
  The change in sleep quality in terms of change in Pittsburgh sleep quality index (PSQI) score
Change in day time sleepiness from the baseline | Baseline, 8 weeks
  The change in daytime sleepiness in terms of change in Epworth sleepiness scale
Change in antioxidant property from the baseline | Baseline, 8 weeks
  The change in antioxidant property in terms of change in serum glutathione reductase
Change in the quality of life from the baseline | Baseline, 8 weeks
  The change in the quality of life in terms of change in Quality of Life in Epilepsy Inventory (QOLIE-31)

CONTACTS AND LOCATIONS:
Overall Officials: Debasish Hota, D.M, Study Chair — AIIMS, Bhubaneswar
Locations (1):
- All India Institute of Medical Sciences (AIIMS), Bhubaneswar, Odisha, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cramer JA, Perrine K, Devinsky O, Bryant-Comstock L, Meador K, Hermann B. Development and cross-cultural translations of a 31-item quality of life in epilepsy inventory. Epilepsia. 1998 Jan;39(1):81-8. doi: 10.1111/j.1528-1157.1998.tb01278.x. PMID 9578017
- [Result] Vimala PV, Bhutada PS, Patel FR. Therapeutic potential of agomelatine in epilepsy and epileptic complications. Med Hypotheses. 2014 Jan;82(1):105-10. doi: 10.1016/j.mehy.2013.11.017. Epub 2013 Nov 21. PMID 24314750
- [Result] Cockerell OC, Sander JW, Shorvon SD. Remission of epilepsy. The NGPS. National General Practice Study of Epilepsy. Lancet. 1995 Nov 4;346(8984):1228. doi: 10.1016/s0140-6736(95)92933-9. No abstract available. PMID 7475682
- [Result] MacDonald BK, Johnson AL, Goodridge DM, Cockerell OC, Sander JW, Shorvon SD. Factors predicting prognosis of epilepsy after presentation with seizures. Ann Neurol. 2000 Dec;48(6):833-41. PMID 11117539
- [Result] Yalyn O, Arman F, Erdogan F, Kula M. A comparison of the circadian rhythms and the levels of melatonin in patients with diurnal and nocturnal complex partial seizures. Epilepsy Behav. 2006 May;8(3):542-6. doi: 10.1016/j.yebeh.2005.12.015. Epub 2006 Mar 9. PMID 16524783
- [Result] Costa-Lotufo LV, Fonteles MM, Lima IS, de Oliveira AA, Nascimento VS, de Bruin VM, Viana GS. Attenuating effects of melatonin on pilocarpine-induced seizures in rats. Comp Biochem Physiol C Toxicol Pharmacol. 2002 Apr;131(4):521-9. doi: 10.1016/s1532-0456(02)00037-6. PMID 11976067
- [Result] Borowicz KK, Kaminski R, Gasior M, Kleinrok Z, Czuczwar SJ. Influence of melatonin upon the protective action of conventional anti-epileptic drugs against maximal electroshock in mice. Eur Neuropsychopharmacol. 1999 Mar;9(3):185-90. doi: 10.1016/s0924-977x(98)00022-4. PMID 10208286
- [Result] Lima E, Cabral FR, Cavalheiro EA, Naffah-Mazzacoratti Mda G, Amado D. Melatonin administration after pilocarpine-induced status epilepticus: a new way to prevent or attenuate postlesion epilepsy? Epilepsy Behav. 2011 Apr;20(4):607-12. doi: 10.1016/j.yebeh.2011.01.018. Epub 2011 Mar 30. PMID 21454134
- [Result] Yahyavi-Firouz-Abadi N, Tahsili-Fahadan P, Riazi K, Ghahremani MH, Dehpour AR. Involvement of nitric oxide pathway in the acute anticonvulsant effect of melatonin in mice. Epilepsy Res. 2006 Feb;68(2):103-13. doi: 10.1016/j.eplepsyres.2005.09.057. Epub 2006 Jan 10. PMID 16406488
- [Result] Goldberg-Stern H, Oren H, Peled N, Garty BZ. Effect of melatonin on seizure frequency in intractable epilepsy: a pilot study. J Child Neurol. 2012 Dec;27(12):1524-8. doi: 10.1177/0883073811435916. Epub 2012 Feb 28. PMID 22378657
- [Result] Gupta M, Aneja S, Kohli K. Add-on melatonin improves quality of life in epileptic children on valproate monotherapy: a randomized, double-blind, placebo-controlled trial. Epilepsy Behav. 2004 Jun;5(3):316-21. doi: 10.1016/j.yebeh.2004.01.012. PMID 15145300
- [Result] Singer MA. Effects of furosemide and ethacrynic acid on cation transport across phospholipid bilayer membranes. Can J Physiol Pharmacol. 1974 Oct;52(5):930-41. doi: 10.1139/y74-122. No abstract available. PMID 4425994
- [Result] Gupta M, Aneja S, Kohli K. Add-on melatonin improves sleep behavior in children with epilepsy: randomized, double-blind, placebo-controlled trial. J Child Neurol. 2005 Feb;20(2):112-5. doi: 10.1177/08830738050200020501. PMID 15794175
- [Result] Gupta M, Gupta YK, Agarwal S, Aneja S, Kohli K. A randomized, double-blind, placebo controlled trial of melatonin add-on therapy in epileptic children on valproate monotherapy: effect on glutathione peroxidase and glutathione reductase enzymes. Br J Clin Pharmacol. 2004 Nov;58(5):542-7. doi: 10.1111/j.1365-2125.2004.02210.x. PMID 15521903
- [Result] Bertaina-Anglade V, Drieu-La-Rochelle C, Mocaer E, Seguin L. Memory facilitating effects of agomelatine in the novel object recognition memory paradigm in the rat. Pharmacol Biochem Behav. 2011 Jun;98(4):511-7. doi: 10.1016/j.pbb.2011.02.015. Epub 2011 Feb 22. PMID 21352847
- [Result] Lopes MC, Quera-Salva MA, Guilleminault C. Non-REM sleep instability in patients with major depressive disorder: subjective improvement and improvement of non-REM sleep instability with treatment (Agomelatine). Sleep Med. 2007 Dec;9(1):33-41. doi: 10.1016/j.sleep.2007.01.011. Epub 2007 Sep 7. PMID 17826314
- [Result] AlAhmed S, Herbert J. Effect of agomelatine and its interaction with the daily corticosterone rhythm on progenitor cell proliferation in the dentate gyrus of the adult rat. Neuropharmacology. 2010 Nov;59(6):375-9. doi: 10.1016/j.neuropharm.2010.05.008. Epub 2010 Jun 1. PMID 20685215
- [Result] Bourin M, Mocaer E, Porsolt R. Antidepressant-like activity of S 20098 (agomelatine) in the forced swimming test in rodents: involvement of melatonin and serotonin receptors. J Psychiatry Neurosci. 2004 Mar;29(2):126-33. PMID 15069466
- [Result] Amudhan S, Gururaj G, Satishchandra P. Epilepsy in India I: Epidemiology and public health. Ann Indian Acad Neurol. 2015 Jul-Sep;18(3):263-77. doi: 10.4103/0972-2327.160093. PMID 26425001
- [Result] Fisher RS, Cross JH, D'Souza C, French JA, Haut SR, Higurashi N, Hirsch E, Jansen FE, Lagae L, Moshe SL, Peltola J, Roulet Perez E, Scheffer IE, Schulze-Bonhage A, Somerville E, Sperling M, Yacubian EM, Zuberi SM. Instruction manual for the ILAE 2017 operational classification of seizure types. Epilepsia. 2017 Apr;58(4):531-542. doi: 10.1111/epi.13671. Epub 2017 Mar 8. PMID 28276064
- [Result] Liu J, Clough SJ, Hutchinson AJ, Adamah-Biassi EB, Popovska-Gorevski M, Dubocovich ML. MT1 and MT2 Melatonin Receptors: A Therapeutic Perspective. Annu Rev Pharmacol Toxicol. 2016;56:361-83. doi: 10.1146/annurev-pharmtox-010814-124742. Epub 2015 Oct 23. PMID 26514204
- [Result] Sanchez-Barcelo EJ, Rueda N, Mediavilla MD, Martinez-Cue C, Reiter RJ. Clinical Uses of Melatonin in Neurological Diseases and Mental and Behavioural Disorders. Curr Med Chem. 2017 Nov 20;24(35):3851-3878. doi: 10.2174/0929867324666170718105557. PMID 28721826
- [Result] Tchekalarova J, Petkova Z, Pechlivanova D, Moyanova S, Kortenska L, Mitreva R, Lozanov V, Atanasova D, Lazarov N, Stoynev A. Prophylactic treatment with melatonin after status epilepticus: effects on epileptogenesis, neuronal damage, and behavioral changes in a kainate model of temporal lobe epilepsy. Epilepsy Behav. 2013 Apr;27(1):174-87. doi: 10.1016/j.yebeh.2013.01.009. Epub 2013 Feb 28. PMID 23435277
- [Result] Mevissen M, Ebert U. Anticonvulsant effects of melatonin in amygdala-kindled rats. Neurosci Lett. 1998 Nov 20;257(1):13-6. doi: 10.1016/s0304-3940(98)00790-3. PMID 9857954
- [Result] Rocha AKAA, de Lima E, Amaral F, Peres R, Cipolla-Neto J, Amado D. Altered MT1 and MT2 melatonin receptors expression in the hippocampus of pilocarpine-induced epileptic rats. Epilepsy Behav. 2017 Jun;71(Pt A):23-34. doi: 10.1016/j.yebeh.2017.01.020. Epub 2017 Apr 28. PMID 28460319
- [Result] Ma Y, Sun X, Li J, Jia R, Yuan F, Wei D, Jiang W. Melatonin Alleviates the Epilepsy-Associated Impairments in Hippocampal LTP and Spatial Learning Through Rescue of Surface GluR2 Expression at Hippocampal CA1 Synapses. Neurochem Res. 2017 May;42(5):1438-1448. doi: 10.1007/s11064-017-2200-5. Epub 2017 Feb 18. PMID 28214985
- [Result] Fenoglio-Simeone K, Mazarati A, Sefidvash-Hockley S, Shin D, Wilke J, Milligan H, Sankar R, Rho JM, Maganti R. Anticonvulsant effects of the selective melatonin receptor agonist ramelteon. Epilepsy Behav. 2009 Sep;16(1):52-7. doi: 10.1016/j.yebeh.2009.07.022. Epub 2009 Aug 13. PMID 19682955
- [Result] Brigo F, Igwe SC, Del Felice A. Melatonin as add-on treatment for epilepsy. Cochrane Database Syst Rev. 2016 Aug 11;2016(8):CD006967. doi: 10.1002/14651858.CD006967.pub4. PMID 27513702
- [Result] Aguiar CC, Almeida AB, Araujo PV, Vasconcelos GS, Chaves EM, do Vale OC, Macedo DS, de Sousa FC, Viana GS, Vasconcelos SM. Anticonvulsant effects of agomelatine in mice. Epilepsy Behav. 2012 Jul;24(3):324-8. doi: 10.1016/j.yebeh.2012.04.134. Epub 2012 Jun 2. PMID 22658946
- [Result] O'Donoghue MF, Duncan JS, Sander JW. The National Hospital Seizure Severity Scale: a further development of the Chalfont Seizure Severity Scale. Epilepsia. 1996 Jun;37(6):563-71. doi: 10.1111/j.1528-1157.1996.tb00610.x. PMID 8641234
- [Result] Buysse DJ, Reynolds CF 3rd, Monk TH, Hoch CC, Yeager AL, Kupfer DJ. Quantification of subjective sleep quality in healthy elderly men and women using the Pittsburgh Sleep Quality Index (PSQI). Sleep. 1991 Aug;14(4):331-8. PMID 1947597
- [Result] Lerche H, Daniluk J, Lotay N, DeRossett S, Edwards S, Brandt C. Efficacy and safety of ezogabine/retigabine as adjunctive therapy to specified single antiepileptic medications in an open-label study of adults with partial-onset seizures. Seizure. 2015 Aug;30:93-100. doi: 10.1016/j.seizure.2015.06.002. Epub 2015 Jun 8. PMID 26216692